CLINICAL TRIAL: NCT03928691
Title: Impact of Body Mass Index on Serum Maternal and Fetal Magnesium Level in Pregnant Recipients of Magnesium Sulphate
Brief Title: Impact of Body Mass Index on Serum Maternal and Fetal Magnesium Level
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Principal investigator, Assiut University
Other Study IDs: MAGPET
Record Dates: First submitted 2019-04-24; First posted 2019-04-26 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Magnesium Sulfate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: pregnant women admitted to Women's Health Hospital , Assiut university during 2019-2020 will be counseled to participate in the study
  Interventions: Drug: Magnesium Sulfate

INTERVENTIONS:
Drug: Magnesium Sulfate — 4 gram MgSo4 diluted in 150 cc saline infused IV within 30 minutes as loading dose then the patient will receive the maintenance dose of 1gram MgSo4 per hour for 6 hours.

SUMMARY:
Magnesium sulphate is an inorganic salt with multiple therapeutic applications in medicine it has been widely utilized and studied on a diverse set of conditions such as asthma, cardiac arrhythmia and stroke. In pregnant women ,MgSo4 has been used in many cases such as for seizures prophylaxis in preeclampsia, tocolysis in preterm labour and for fetal neuroprotection in immenint preterm delivery.MgSo4 has been used as the standard drug for tocolysis in preterm labour and other drugs have been compared to it.

ELIGIBILITY:
Inclusion criteria:

pregnant women 34 weeks or less admitted to Women's Health Hospital with a diagnosis of :

* sever preeclampsia. It is defined as 1- blood pressure 160/110 mmHg or more 2- proteinurea (+3 or more by dipstick) 3-HELLP syndrome
* threatened preterm labour that will receive Magnesium Sulphate either for tocolysis or neuroprotection.

Exclusion criteria:

- women with more than 34 weeks gestation and with any contraindication for Magnesium Sulphate intake like severe renal impairment or myasthenia gravis.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: women included will be classified according to BMI underwieght ( less than 18.85) , Normal weight (18.5-24.9)
  , Overweight (25-29.9) and obese (30 or more)
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-06-30 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
the percentage of women reaching the Mg therapeutic level. | 24 hours
  the Mg therapeutic level of 4,8 mg/dl.

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No